CLINICAL TRIAL: NCT01250600
Title: Application of Intelligent Wireless and Portable Tele-Cardiopulmonary Exercise System on Rehabilitation for Patients With Myocardial Infarction
Brief Title: Effects of Intelligent Tele-Cardiopulmonary Exercise System on Rehabilitation for Patients With Myocardial Infarction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China Medical University Hospital (Other)
Collaborators: China Medical University, China (Other)
Responsible Party: Nai-Hsin Meng, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMU99-NCTU-12
Record Dates: First submitted 2010-11-26; First posted 2010-12-01 (Estimated); Last update posted 2010-12-01 (Estimated); Status verified 2010-11

CONDITIONS: Exercise Capacity

ARMS (2):
- Remote-care (Experimental): Home exercise monitored by the remote care system
  Interventions: Behavioral: Home exercise
- Control (Active Comparator): Home exercise under expert's instruction
  Interventions: Behavioral: Home exercise

INTERVENTIONS:
Behavioral: Home exercise — Daily home exercise for 3 months

SUMMARY:
Although a lot of evidence and guidelines recommend that patients have cardiac rehabilitation, in reality, the actual rate cardiac patients entering cardiac rehabilitation program is low, usually less than one third. One of the main hindrances of patients participating cardiac rehabilitation program is insufficient number of medical institutions that can provide rehabilitation services. Patients usually cannot perform exercise program under medical professionals monitoring without having to go far. This spatial and temporal difficulty led to the low rate of patients taking cardiac rehabilitation program. The risk of patients to do exercise is higher than healthy adult.

This project will develop the intelligent portable remote care system for cardiopulmonary exercise to provide an instant ECG monitoring service through the integration of front-end wireless ECG measuring devices, expert system, and back-end tele-care platform. Many patients are inconvenient to go to large hospital regularly for cardiac rehabilitation training. This project will help them to exercise at home after once or twice rehabilitation training in clinic for each month and the medical professional will supervise remotely to see how much exercise they did. For that reason the project can help to break through spatial and temporal difficulty of having cardiac rehabilitation, so that cardiac rehabilitation can be help more patients. Patients have this tele-care system while they are doing exercise at home, the built-in heart rate and cardiac rhythm warning function will remind them to take a break, even to take medical treatment. More importantly, the ECG signal can be almost immediately (real time) uploaded by network to the chest pain unit of hospital. The cardiology expert will be aware of the warning at the first moment. This is an important protection to patients' safety of doing rehabilitation sports at home.

This randomized control trial will recruit 80 patients who had myocardial infarction within 6 weeks, and are not able to attend a hospital based cardiac rehabilitation program regularly. All patient will undergo a three-month home exercise program under the instruction provided by the physiatrists and physiotherapists. Forty of them (the remote-care group) will use the intelligent portable remote care system for cardiopulmonary exercise to monitor their exercise intensity and cardiac rhythm during exercise. The other 40 patients (the control group) undertake the exercise program at home without using the remote care system. The efficacy and safety of exercise program will be compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* within 6 weeks after an acute myocardial infarction
* not able to attend a hospital based cardiac rehabilitation program regularly

Exclusion Criteria:

* with left ventricular ejection fraction lower than 40%
* history of cardiac arrest
* history of cardiogenic shock, heart failure
* complicated arrhythmia
* abnormal exercise hemodynamics: blood pressure not increased with exercise
* any other physical/psychological condition that hinders the patient's walking ability

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-12 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in exercise capacity at 3 months | baseline and after a 3-month exercise program
  6-minute walk test and maximum oxygen uptake obtained by a graded exercise test

SECONDARY OUTCOMES:
Change from baseline in quality of life at 3 months. | baseline and after a 3-month exercise program
  Quality of life questionnaires, including SF-36
Change from baseline in physical activities at 3 months. | baseline and after a 3-month exercise program
  The International Physical Activity Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Nai-Hsin Meng, M.D., Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan, Taiwan